CLINICAL TRIAL: NCT04093596
Title: A Single-Arm, Open-Label, Phase 1 Study of the Safety, Efficacy, and Cellular Kinetics/Pharmacodynamics of ALLO-715 to Evaluate an Anti-BCMA Allogeneic CAR T Cell Therapy With or Without Nirogacestat in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: Safety and Efficacy of ALLO-715 BCMA Allogenic CAR T Cells in in Adults With Relapsed or Refractory Multiple Myeloma (UNIVERSAL)
Acronym: UNIVERSAL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Allogene Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-715-101
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine; Cyclophosphamide; nirogacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALLO-647, ALLO-715, Nirogacestat (Experimental)
  Interventions: Genetic: ALLO-715; Biological: ALLO-647; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Nirogacestat

INTERVENTIONS:
Genetic: ALLO-715 — ALLO-715 is an allogeneic CAR T cell therapy targeting BCMA
Biological: ALLO-647 — ALLO-647 is a monoclonal antibody that recognizes a CD52 antigen
Drug: Fludarabine — Chemotherapy for lymphodepletion
Drug: Cyclophosphamide — Chemotherapy for lymphodepletion
Drug: Nirogacestat — a small molecule, selective, reversible, noncompetitive inhibitor of γsecretase (GSI) that increases BCMA target density on the surface of multiple myeloma cells.

SUMMARY:
The purpose of the UNIVERSAL study is to assess the safety, efficacy, cell kinetics, and immunogenicity of ALLO-715 with or without Nirogacestat in adults with relapsed or refractory multiple myeloma after a lymphodepletion regimen of ALLO-647 in combination with fludarabine and/or cyclophosphamide, or ALLO-647 alone.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of relapsed/refractory multiple myeloma (MM) with measurable disease (serum, urine, or free light chain [FLC]) per International Myeloma Working Group (IMWG) criteria
* At least 3 prior lines of MM therapy, including a proteasome inhibitor, immunomodulatory agent, and anti-CD38 antibody (unless contraindicated), and refractory to the last treatment line.
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Absence of donor (product)-specific anti-HLA antibodies
* Adequate hematologic, renal, hepatic, pulmonary, and cardiac function

Exclusion Criteria:

* Current or history of Central Nervous System (CNS) involvement of myeloma or plasma cell leukemia
* Clinically significant CNS disorder
* Current or history of thyroid disorder
* Autologous stem cell transplant within the last 6 weeks, or any allogeneic stem cell transplant
* Prior treatment with anti-BCMA therapy, any gene therapy, any genetically modified cell therapy, or adoptive T cell therapy
* History of HIV infection or acute or chronic active hepatitis B or C infection
* Patients unwilling to participate in an extended safety monitoring period

Additional Exclusion Criteria for Nirogacestat plus ALLO-715 Cohorts

* Inability to swallow tablets
* Subject has known malabsorption syndrome or preexisting gastrointestinal conditions that may impair absorption of nirogacestat
* Use of strong/moderate CYP3A4 inhibitors, and strong CYP3A4 inducers within 14 days before starting nirogacestat.
* Use of concomitant medications that are known to prolong the QT/QTcF interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects experiencing Dose Limiting Toxicities at increasing doses of ALLO-715 | 28 Days
  Dose limiting toxicities are defined as ALLO-715-related adverse events with onset within 28 days following infusion of ALLO-715.
To assess the overall safety profile and tolerability of ALLO-647 in combination with Fludarabine and/or cyclophosphamide or ALLO-647 alone, prior to ALLO-715 to confirm the dose of ALLO-647. | 33 days
  The proportion of subjects in a dose cohort with DLTs of ALLO-647
To assess the overall safety profile and tolerability of nirogacestat given concomitantly with ALLO-715 following lymphodepletion with Flu/ Cy/ ALLO-647. | 28 days
  Dose limiting toxicities are defined as ALLO-715-related adverse events with onset within 28 days following infusion of ALLO-715.

SECONDARY OUTCOMES:
Cellular kinetics of ALLO-715 | up to 60 months
  Levels of anti-BCMA CAR T cells in blood
antitumor activity of ALLO-715 in combination with nirogacestat | up to 60 months
  overall -response rate (ORR)
Cellular kinetics of ALLO-715 in combination with nirogacestat | up to 60 months
  Levels of anti-BCMA CAR T cells in blood
Pharmacokinetics of ALLO-647 | up to 60 months
  Serum concentration levels of ALLO-647
Pharmacokinetics of nirogacestat | up to 60 months
  Serum concentration levels of nirogacestat
Incidence of immunogenicity against ALLO-715 and ALLO-647 | up to 60 months
  detection and levels of anti-drug antibodies
Immune monitoring after lymphodepletion regimen | up to 60 months
  Detection of the following circulating cells: T cell subset, B lymphocytes, and NK cells
Anti-tumor activity of ALLO-715 | up to 60 months
  overall response rate
Anti-tumor activity of ALLO-715 | up to 60 months
  duration of response
Anti-tumor activity of ALLO-715 | up to 60 months
  overall survival
Anti-tumor activity of ALLO-715 | up to 60 months
  minimal residual disease
To evaluate the expression of BCMA in bone marrow plasma cells with and without nirogacestat | up to 60 months
  Overall response rate of ALLO-715 with and without Nirogacestat

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - Stanford Cancer Institute, Palo Alto, California
  - Sarah Cannon/Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Mailankody S, Matous JV, Chhabra S, Liedtke M, Sidana S, Oluwole OO, Malik S, Nath R, Anwer F, Cruz JC, Htut M, Karski EE, Lovelace W, Dillon M, Butz E, Ying W, Balakumaran A, Kumar SK. Allogeneic BCMA-targeting CAR T cells in relapsed/refractory multiple myeloma: phase 1 UNIVERSAL trial interim results. Nat Med. 2023 Feb;29(2):422-429. doi: 10.1038/s41591-022-02182-7. Epub 2023 Jan 23. PMID 36690811
- [Derived] Abba Moussa D, Vazquez M, Chable-Bessia C, Roux-Portalez V, Tamagnini E, Pedotti M, Simonelli L, Ngo G, Souchard M, Lyonnais S, Chentouf M, Gros N, Marsile-Medun S, Dinter H, Pugniere M, Martineau P, Varani L, Juan M, Calderon H, Naranjo-Gomez M, Pelegrin M. Discovery of a pan anti-SARS-CoV-2 monoclonal antibody with highly efficient infected cell killing capacity for novel immunotherapeutic approaches. Emerg Microbes Infect. 2025 Dec;14(1):2432345. doi: 10.1080/22221751.2024.2432345. Epub 2024 Dec 9. PMID 39584380